CLINICAL TRIAL: NCT06235749
Title: Administration Of Calcium Gluconate for The Reduction of Blood Loss During Elective Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RMB-0605-22
Record Dates: First submitted 2023-11-20; First posted 2024-02-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Elective Cesarean Delivery
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- calcium gluconate (Experimental): Administration of Calcium Gluconate 10% IV following umbilical cord clamping.
  Interventions: Drug: Calcium Gluconate 10%
- normal saline 0.9% (Placebo Comparator): Administration of normal saline 0.9% IV following umbilical cord clamping.
  Interventions: Drug: sodium chloride 0.9%

INTERVENTIONS:
Drug: Calcium Gluconate 10% — Administration of Calcium Gluconate 10% IV following umbilical cord clamping
  Arms: calcium gluconate
Drug: sodium chloride 0.9% — Administration of sodium chloride 0.9% IV following umbilical cord clamping
  Arms: normal saline 0.9%

SUMMARY:
Postpartum hemorrhage (PPH) is the leading cause of death related to pregnancy. PPH can lead to blood transfusion, disseminated intravascular coagulation (DIC), hysterectomy, or death. The prophylactic administration of uterotonic agents as part of an active management of the third stage of labor has been proven to reduce rates of PPH. However, even with these treatments, PPH rate is still relatively high, and puts women at risk of heavy bleeding and death.

Calcium is a key component in the coagulation cascade and known as factor IV. It has a role in platelet activation, and it is an important co-factor for the activation of factors II and There is a concentration-dependent effect of hypocalcemia on in vitro clot strength in patients at risk of bleeding. Calcium gluconate is the calcium salt of gluconic acid, and it has a relatively strong safety profile.

Hypocalcemia is a poor prognostic factor in actively bleeding patients. Calcium has a positive inotropic effect both on skeletal muscle and smooth muscle. The inotropic effect doesn't skip the myometrium, and it is well-established that hypocalcemia can impair myometrial contractility. As so, calcium channel blockers are prescribed as a tocolytic drug and calcium gluconate should be considered as adjuvant therapy for treating PPH duo to atony, in case of prolonged tocolytic or magnesium sulfate use prior to delivery. Studies have already shown an association between low ionized calcium levels and the risk for severe bleeding. In a pilot randomized controlled trial of patients with risk factors for uterine atony, calcium was shown to reduce uterine atony compared to placebo. However, current studies have small sample size and are limited to a high-risk population. There are no recommendations in current guidelines for monitoring calcium levels or prescribing calcium as a prophylactic measure for the third stage of labor, despite atony and coagulopathy being significant causes of PPH.

HYPOTHESIS: Administration of Calcium Gluconate at the third stage of elective Cesarean delivery will decrease the rates of blood loss during and after the surgery by reducing the rates of uterine atony and development of coagulopathy, thus has the potential of reducing the incidence of PPH and its complications without severe side effects.

DETAILED DESCRIPTION:
After signing a consent form prior to the surgery (at the pre-operative assessment), At the third stage of labor, women who gave their consent to participate in the study will get either 10 ml of Calcium Gluconate 10% solution (containing 0.94 gr of calcium gluconate) diluted in 100 ml of normal saline IV or 110 ml of normal saline IV.

The solutions will be given in addition to Carbetocin (a long acting oxytocin analogue), in both arms. The invastigators will use calcium gluconate during even-numbered months and normal saline during odd-numbered months, or vice versa, according to randomization that will be known to the primary researcher alone.

A blood sample will be drawn at the beginning of the surgery and sent for blood gas analysis, determining ionized calcium levels and coagulation profile. Women with hypocalcemia or hypercalcemia will be excluded from the trial. Only patients with normal calcium levels between 1.0-1.3 mmol/L will be included in this trial.

An ECG strip will be done prior to the surgery, making sure that the patient doesn't suffer from a QT segment abnormality. All patients will be monitored with a 3 lead- ECG prior, during, and 2 hours following calcium administration. Patients with QT interval abnormalities will be excluded from the trial. After the surgery, a blood sample will be drawn and sent to blood gas analysis (determining ionized calcium levels) and for coagulation profile. A complete blood count will be routinely taken for all women the next day. The hemoglobin level will be compared to the hemoglobin level prior to CD.

Decreased mean hemoglobin drop is the primary outcome. the secondary outcomes are described below.

After the primary analysis we will perform a subgroup analysis, determine whether women with high risk for PPH (such as overdistended uterus, abnormal placentation, myomatous uterus, grand multiparty, coagulation disorder, etc.) may benefit from the intervention more than the general population of all participants.

ELIGIBILITY:
Inclusion Criteria:

- Elective Cesarean Delivery, at Gestational age of 35 weeks or more.

Exclusion Criteria:

* Age younger than 18 years old.
* Patients treated with calcium channel blockers.
* Chronic renal failure and hyperphosphatemia.
* Sarcoidosis.
* Hypocalcemia (ionized Ca<1 mmol/L) or hypercalcemia (ionized Ca> 1.3 mmol/L) before the surgery.
* Any QT abnormalities as evident by ECG before Calcium Gluconate administrations or any known conduction abnormality.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1180 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean hemoglobin drop | 24 hours after the surgery
  Change in mean hemoglobin drop after cesarean delivery at the Calcium gluconate arm, compared to the control arm.

SECONDARY OUTCOMES:
The rate of women with a decrease of hemoglobin levels of 2 gr/dl or more | 24 hours after the surgery
  The rate of women with a decrease of hemoglobin levels of 2 gr/dl or more.
additional therapy for the management of PPH | during hospitalization, an average of 4 days
  additional therapy for the management of PPH
Receipt of blood products. | during hospitalization, an average of 4 days
  Receipt of blood products.
treatment with intravenous ferrous (iron). | during hospitalization, an average of 4 days
  treatment with intravenous ferrous (iron).
estimated blood loss during the surgery. | during the surgery
  estimated blood loss during the surgery.
Hospitalization length of stay. | an average of 4 days
  Hospitalization length of stay.
Duration of cesarean delivery | during the surgery
  Duration of cesarean delivery
A composite of adverse maternal outcomes | during hospitalization, an average of 4 days
  A composite of adverse maternal outcomes including at least one of the following: admission to intensive care unit (NICU), the need for a surgical treatment for uncontrolled PPH, massive blood transfusion (defined as transfusion of ≥10 units red blood cells (RBCs) in 24 hours, disseminated intravascular coagulation (DIC), and death.
Endometritis or antibiotic treatment following CD. | during hospitalization, an average of 4 days
  Endometritis or antibiotic treatment following CD.

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Shamir Medical Center, Be’er Ya‘aqov
  - Rambam Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deneux-Tharaux C, Bonnet MP, Tort J. [Epidemiology of post-partum haemorrhage]. J Gynecol Obstet Biol Reprod (Paris). 2014 Dec;43(10):936-50. doi: 10.1016/j.jgyn.2014.09.023. Epub 2014 Nov 6. French. PMID 25447386
- [Background] Palta S, Saroa R, Palta A. Overview of the coagulation system. Indian J Anaesth. 2014 Sep;58(5):515-23. doi: 10.4103/0019-5049.144643. PMID 25535411
- [Background] Ho KM, Yip CB. Concentration-dependent effect of hypocalcaemia on in vitro clot strength in patients at risk of bleeding: a retrospective cohort study. Transfus Med. 2016 Feb;26(1):57-62. doi: 10.1111/tme.12272. Epub 2016 Jan 5. PMID 26729371
- [Background] Papandreou L, Chasiotis G, Seferiadis K, Thanasoulias NC, Dousias V, Tsanadis G, Stefos T. Calcium levels during the initiation of labor. Eur J Obstet Gynecol Reprod Biol. 2004 Jul 15;115(1):17-22. doi: 10.1016/j.ejogrb.2003.11.032. PMID 15223159
- [Background] Korytny A, Klein A, Marcusohn E, Freund Y, Neuberger A, Raz A, Miller A, Epstein D. Hypocalcemia is associated with adverse clinical course in patients with upper gastrointestinal bleeding. Intern Emerg Med. 2021 Oct;16(7):1813-1822. doi: 10.1007/s11739-021-02671-6. Epub 2021 Mar 2. PMID 33651325
- [Background] Epstein D, Freund Y, Marcusohn E, Diab T, Klein E, Raz A, Neuberger A, Miller A. Association Between Ionized Calcium Level and Neurological Outcome in Endovascularly Treated Patients with Spontaneous Subarachnoid Hemorrhage: A Retrospective Cohort Study. Neurocrit Care. 2021 Dec;35(3):723-737. doi: 10.1007/s12028-021-01214-3. Epub 2021 Apr 7. PMID 33829378
- [Background] Kawarabayashi T, Kishikawa T, Sugimori H. Effects of external calcium, magnesium, and temperature on spontaneous contractions of pregnant human myometrium. Biol Reprod. 1989 May;40(5):942-8. doi: 10.1095/biolreprod40.5.942. PMID 2765618
- [Background] Epstein D, Solomon N, Korytny A, Marcusohn E, Freund Y, Avrahami R, Neuberger A, Raz A, Miller A. Association between ionised calcium and severity of postpartum haemorrhage: a retrospective cohort study. Br J Anaesth. 2021 May;126(5):1022-1028. doi: 10.1016/j.bja.2020.11.020. Epub 2020 Dec 17. PMID 33341222
- [Background] Ansari JR, Kalariya N, Carvalho B, Flood P, Guo N, Riley E. Calcium chloride for the prevention of uterine atony during cesarean delivery: A pilot randomized controlled trial and pharmacokinetic study. J Clin Anesth. 2022 Sep;80:110796. doi: 10.1016/j.jclinane.2022.110796. Epub 2022 Apr 18. PMID 35447502

DOCUMENTS (1):
  • Study Protocol (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT06235749/Prot_000.pdf